CLINICAL TRIAL: NCT04353622
Title: Exoskeleton-assisted Upper Limb Rehabilitation After Stroke: A Randomized Controlled Trial
Brief Title: Exoskeleton-assisted Upper Limb Rehabilitation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, iremakgun, Physiotherapist, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09.2019.146
Record Dates: First submitted 2020-02-21; First posted 2020-04-20 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Stroke; Upper Extremity Dysfunction
Keywords: Stroke; Upper extremity; Robotic rehabilitation; Motor function; Quality of life
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted Treatment (Active Comparator): Rehabilitation protocol was applied with robotic device (HOUSTONBIONİCS ExoRehab UE1).
  Interventions: Device: Exoskeleton robot for upper extremity
- Conventional Physiotherapy (Active Comparator): Conventional physiotherapy program included neurophysiological approaches.
  Interventions: Other: Conventional physiotherapy

INTERVENTIONS:
Device: Exoskeleton robot for upper extremity — Robot-assisted Treatment Program:
  * 10 minutes elbow flexion/extension
  * 10 minutes forearm supination/pronation
  * 10 minutes wrist flexion/extension
  * 10 minutes ulnar/radial deviation
  Frequency: 2/week Duration: 12 sessions (6 weeks)
  Arms: Robot-assisted Treatment
Other: Conventional physiotherapy — Ferquency: 2/week Duration: 12 sessions (6weeks) Each session: 50 minutes
  Arms: Conventional Physiotherapy

SUMMARY:
In recent studies, it has been observed that robotic devices make a positive contribution to motor recovery and the activities of daily living. However, studies about the effects of stroke rehabilitation with robotic devices are limited.

This study aimed to investigate the effect of upper extremity robotic rehabilitation on motor function and quality of life in stroke patients.

DETAILED DESCRIPTION:
Stroke survivors have difficulties in participating in activities of daily living due to functional disabilities. The majority of patients after stroke need rehabilitation to gain independence in daily life as the first target. Therefore, different treatment approaches are used in stroke rehabilitation.

The use of technology in stroke rehabilitation has become very common in recent years. Robotic devices used in rehabilitation enhance the healing process by giving patients more intensive and task-oriented exercises. A lot of systematic and meta-analysis studies have shown that robot-assisted devices provide positive motor recoveries, especially in the treatment of upper extremities. However, the optimal timing, duration, and dose of robotic rehabilitation that should be applied after stroke remain uncertain.

In the light of this information, this study examines the effects of the robotic device produced for upper limb rehabilitation on daily life activities and motor function.

ELIGIBILITY:
Inclusion Criteria:

* Having ischemic or hemorrhagic stroke history
* Being at the age between 40 and 85
* MAS (Modified Ashworth Scale) < 3 for upper extremity
* At least 6 months after stroke
* Participants who agree to participate in the study

Exclusion Criteria:

* Cardiovascular weakness (severe hypertension, coronary artery disease)
* Mini-Mental State Examination score < 24
* Recurrent stroke
* Having other orthopedic and neurologic conditions that may affect upper extremity movement
* Having behavioral and cognitive problems

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 24 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Upper Extremity Assessment | before treatment and at six weeks of the beginning of the treatment
  Fugl-Meyer Upper Extremity Assessment is an index to assess physical performance in individuals who had a stroke. This index consists of 33 items. Each item scored between 0 and 2. The highest score for the upper extremity is 66.
Modified Ashworth Scale | before treatment and at six weeks of the beginning of the treatment
  Modified Ashworth Scale is used for measuring the spasticity of upper extremity skeletal muscle. The Modified Ashworth Scale (MAS) is scored from 0 to 5 to measure the resistance encountered when performing passive muscle stretching. The lowest score is 0 (no spasticity) and the highest score is 5 (severe spasticity).

SECONDARY OUTCOMES:
Upper Extremity Motor Activity Log | before treatment and at six weeks of the beginning of the treatment
  Upper Extremity Motor Activity Log consists of two subscales (amount of use and quality of movement) that determine how often the patient uses the affected side in daily life activities and how successful this activity is. Items on each scale are scored between 0 and 5.
Nottingham Extended Activities of Daily Living Scale | before treatment and at six weeks of the beginning of the treatment
  Nottingham Extended Activities of Daily Living Scale is designed for stroke patients but can be also used for other diseases. The scale has 22 items divided into 4 areas of daily life. These areas are mobility, kitchen, domestic and leisure activities. Each item scored between 0 and 3. The highest score of scale is 66.

OTHER OUTCOMES:
Mini-Mental State Examination | Before treatment
  Mini-Mental State Examination is used to determine the cognitive level. This scale consists of 11 items. The highest score is 30. 24 and higher scores are considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: İrem Akgün, Principal Investigator — Marmara University
Locations (1):
- Marmara University Faculty of Health Sciences, Istanbul, Turkey (Türkiye)